CLINICAL TRIAL: NCT06498310
Title: Multicenter Retrospective Cohort Study on Invasive Fungal Infections With Filamentous Fungi in Heart Transplant Patients
Brief Title: Retrospective Study of Invasive Fungal Infections With Filamentous Fungi in Heart Transplant Patients
Acronym: IMI-CART
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9066
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Invasive Fungal Infections
Keywords: Invasive Fungal Infections; Filamentous fungi; Heart transplant; Fungal infections
MeSH Terms: conditions — Invasive Fungal Infections; Mycoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Invasive filamentous fungal infections (aspergillosis, scedosporiosis, mucormycosis, fusarium wilt) are common and serious in immunocompromised subjects and particularly organ transplant patients. There is little recent data in heart transplantation, particularly on the incidence and risk factors of fungal infections. . It is therefore important to have recent data on incidence, risk and prognostic factors in order to improve the management of this severe complication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥18 years old
* Heart transplant
* Invasive fungal infection with filamentous fungi during the period from January 1, 2008 to December 31, 2022
* Proven or probable infection with filamentous fungi according to EORTC/MSGERC criteria (20):

  * Invasive aspergillosis
  * Mucormycosis
  * Fusarium wilt
  * Scedosporiosis
  * Other filamentous fungus infection
* Subject who has not expressed, after information, his opposition to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Patient having expressed his opposition to participating in the study
* Patient not having a liver transplant
* Subject under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient ≥18 years old having heart transplant and invasive fungal infection with filamentous fungi during the period from January 1, 2008 to December 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
To identify the incidence, risk factors and prognostic factors associated with invasive fungal infections caused by filamentous fungi in heart transplant patients. | Up to 2 years
  1. Incidence: number of cases of invasive fungal infection compared to the number of heart transplant patients per year in the study centers
  2. Risk factors: Case-control study. Clinical, microbiological or radiological factors statistically associated with cases of invasive fungal infection compared to controls.
  3. Prognostic factors: Clinical, microbiological or radiological factors of invasive fungal infections associated with mortality at the 12th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France